CLINICAL TRIAL: NCT06787898
Title: USG-Guided Retrolaminar Block Improves Postoperative Gastrointestinal System Functions in Percutaneous Nephrolithotomy Patients: A Prospective, Randomised, Clinical Study
Brief Title: Retrolaminar Block Improves Postoperative Gastrointestinal System Functions:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Principal Investigator, Serpil Bayındır, Principal Investigator, Elazıg Fethi Sekin Sehir Hastanesi
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: FSCH-SB-2024/12-14
Record Dates: First submitted 2024-12-22; First posted 2025-01-22 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Retrolaminar Block; Percutaneous Nephrolithotomy (PCNL)
Keywords: Percutaneous nephrolithotomy; Retrolaminar block

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group R ( The group of patients who underwent retrolaminar block for analgesia) (Other): Retrolaminar block is a simple and easy to perform paravertebral block. Place of application Intraoperative and postoperative analgesia is achieved by applying local anaesthetic between the lamina of the arcus vertebrae and paraspinous muscles under ultrasound guidance.
  Interventions: Other: Group R: retrolaminar block performed group
- Group C (Other): Group C control group without local anaesthetic and block
  Interventions: Other: Group C - Placebo

INTERVENTIONS:
Other: Group R: retrolaminar block performed group — Patients were placed on their side and then T9, T10 vertebrae were marked. After the skin was cleaned and the area was covered with sterile drape. A linear ultrasound probe (6-13 Hz, Hitachi Europe Ltd, Tokyo, Japan) was placed in the middle of the vertebral bodies to image the T9, T10 vertebraes. An experienced anaesthesiologist in RLB performed the procedures with a USG-guided 1-15 Hz convex probe (8-4, Hitachi Europe Ltd, Tokyo, Japan) by in-plane approach. A puncture needle (21Gx100mm, USG-Type CCR, Vygon Co. Ltd. Ecouen, France) was inserted 1 cm from the probe at a 45-degree angle to the skin, targeting the lamina of the desired vertebra. The needle was gently withdrawn to ensure that no blood or cerebrospinal fluid was present. 10 mL of 0.25% bupivacaine (Bupivon®) was injected posterior to each lamina (T9, T10), totalling 20 mL
  Arms: Group R ( The group of patients who underwent retrolaminar block for analgesia)
Other: Group C - Placebo — Patients were placed on their side and then T9, T10 vertebrae were marked. After the skin was cleaned and the area was covered with sterile drape. A linear ultrasound probe (6-13 Hz, Hitachi Europe Ltd, Tokyo, Japan) was placed in the middle of the vertebral bodies to image the T9, T10 vertebraes. An experienced anaesthesiologist in RLB performed the procedures with a USG-guided 1-15 Hz convex probe (8-4, Hitachi Europe Ltd, Tokyo, Japan) by in-plane approach. A puncture needle (21Gx100mm, USG-Type CCR, Vygon Co. Ltd. Ecouen, France) was inserted 1 cm from the probe at a 45-degree angle to the skin, targeting the lamina of the desired vertebra. The needle was gently withdrawn to ensure that no blood or cerebrospinal fluid was present. 10 mL of 0.25% bupivacaine (Bupivon®)was injected posterior to each lamina (T9, T10), totalling 20 mL.
  Arms: Group C

SUMMARY:
Rapid recovery of postoperative bowel function is one of the important goals of accelerated recovery after surgery (ERAS protocols). Gastrointestinal dysfunctions may occur after general anaesthesia. All these lead to a series of adverse outcomes including prolonged hospital stay, high treatment costs and deterioration of patient comfort.

Percutaneous nephrolithotomy (PNL) is the treatment of choice for sizable and intricate kidney stones. Providing effective postoperative pain control is important in preventing respiratory and thromboembolic complications and ensuring patient comfort as well as shortening the hospital stay. The application of USG-guided nerve blocks for analgesia reduces intraoperative opioid use and provides early recovery of postoperative GI dysfunctions. Retrolaminar block (RLB), have been shown to reduce perioperative opioid consumption. Nerve blocks may relieve inflammation-related gastrointestinal dysfunctions by attenuating postoperative inflammatory responses.

This study aimed to determine the effects of USG-guided retrolaminar block on the postoperative gastrointestinal system in patients undergoing PNL.

DETAILED DESCRIPTION:
Rapid recovery of postoperative bowel function is one of the important goals of accelerated recovery after surgery (ERAS protocols). Gastrointestinal dysfunctions such as nausea-vomiting, distension, slowing of intestinal peristalsis, ileus, fatigue, delayed gastric emptying and delayed oral active eating may occur after general anaesthesia. All these lead to a series of adverse outcomes including prolonged hospital stay, high treatment costs and deterioration of patient comfort.

Percutaneous nephrolithotomy (PNL) is the treatment of choice for sizable (>2 cm) and intricate kidney stones. This minimally invasive surgical technique entails the creation of a percutaneous tract through which specialised instruments are inserted to fragment and extract the renal calculi. In the first 24 hours postoperatively, incisional pain is both somatic and visceral in character due to distension in the renal capsule-pelvic- pelvical system and the inserted nephrostomy tube and is carried by the T8-L1 spinal nerves. Blocking the nerves innervating these regions provides an effective analgesia. Providing effective postoperative pain control is important in preventing respiratory and thromboembolic complications and ensuring patient comfort as well as shortening the hospital stay. The application of USG-guided nerve blocks for analgesia reduces intraoperative opioid use and provides early recovery of postoperative GI dysfunctions. Various nerve blocks including retrolaminar block (RLB), erector spina area block (ESPB), and trans abdominal area block (TAPB) have been shown to reduce perioperative opioid consumption. Nerve blocks may relieve inflammation-related gastrointestinal dysfunctions by attenuating postoperative inflammatory responses.

This study aimed to determine the effects of USG-guided retrolaminar block on the postoperative gastrointestinal system in patients undergoing percutaneous nephrolithotomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) I-II-III,
* 18-65 years
* unilateral PNL performed under elective conditions

Exclusion Criteria:

* body mass index > 40 kg/m2,
* inability to understand the pain verbal rating scale and patient-controlled analgesia,
* emergency reoperations,
* ASA 4 or 5,
* drug and alcohol dependence,
* drug allergy,
* Coagulation disorders,
* anatomical abnormalities of the genitourinary system,
* gastrointestinal motility disorders,
* previous abdominal surgery,
* cognitive or psychiatric disorders, mental disorders,
* presence of severe systemic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the detection of gastrointestinal motility disorders (peristaltic activity) in the postoperative period with intermittent USG imaging as a result of decreased opioid consumption during surgery. | Hour 1, Hour 3, Hour 6, and Hour 12 after surgery
  The primary outcome measures were abdominal calculation of Perlas Score (No fluid in the antrum was scored as 0, minimal fluid in the right supine position was scored as 1, and tense antrum in both supine and right supine position was scored as 2) with USG examination after extubation, hour 1, hour 3, hour 6, and hour 12

SECONDARY OUTCOMES:
postoperative gastrointestinal tract function | Hour 1, Hour 3, Hour 6, Hour 12.
  time of first oral feeding, flatus, defecation, mobilisation (min); rescue analgesia time (min) postoperative.
Postoperative analgesia | after extubation, Hour 1, Hour 3 , Hour 6 , and Hour 12.
  VAS Scores (Visual Analog Scale) (In a VAS score of 1-10, each number represents a rough equivalent of the intensity of pain felt. 0: No pain, 10: Intolerable most severe pain)
gastrointestinal tract dysfunction | Hour 1, Hour 3,Hour 6, Hour 12.
  İ-FEED Score values (The I-FEED (intake, nausea sensation, vomiting, physical examination and duration of symptoms) Score was calculated and patients were then categorized into one of three groups: Normal gastrointestinal function score 0-2, postoperative gastrointestinal intolerance (nausea, vomiting or abdominal distension) score 3-5, postoperative ileus score 6-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Elazığ Fethi Sekin City Hospital, Elâzığ, Seçiniz, Turkey (Türkiye)

REFERENCES:
- [Result] Onishi E, Toda N, Kameyama Y, Yamauchi M. Comparison of Clinical Efficacy and Anatomical Investigation between Retrolaminar Block and Erector Spinae Plane Block. Biomed Res Int. 2019 Mar 28;2019:2578396. doi: 10.1155/2019/2578396. eCollection 2019. PMID 31032339
- [Result] Liu D, Xu X, Zhu Y, Liu X, Zhao F, Liang G, Zhu Z. Safety and Efficacy of Ultrasound-Guided Retrolaminar Block of Multiple Injections in Retroperitoneal Laparoscopic Nephrectomy: A Prospective Randomized Controlled Study. J Pain Res. 2021 Feb 5;14:333-342. doi: 10.2147/JPR.S282500. eCollection 2021. PMID 33574697
- See also: pubmed — https://pubmed.ncbi.nlm.nih.gov/33574697/